CLINICAL TRIAL: NCT03676231
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SGM-1019 Administered for 12 Weeks in Subjects With F1-F3 Nonalcoholic Steatohepatitis (NASH)
Brief Title: Study of SGM-1019 in Patients With Nonalcoholic Steatohepatitis (NASH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to a safety event which rendered the risk-benefit profile in NASH to no longer be adequately favorable
Sponsor: Second Genome (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGM-1019-102
Record Dates: First submitted 2018-09-05; First posted 2018-09-18 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High-dose SGM-1019 (Experimental)
  Interventions: Drug: SGM-1019
- Low-dose SGM-1019 (Experimental)
  Interventions: Drug: SGM-1019
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SGM-1019 — Active
  Arms: High-dose SGM-1019; Low-dose SGM-1019
Drug: Placebo — Inactive
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study evaluating the safety, pharmacokinetics, and pharmacodynamics of 12 weeks' administration of SGM-1019 in subjects with fibrosis stage 1-3 (F1-F3) NASH.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 to 75 years, inclusive
* Elevated ALT
* F1-F3 NASH
* BMI ≥ 25

Exclusion Criteria:

* Use of prohibited medication/supplements
* Poorly controlled type 2 diabetes
* Hepatic decompensation
* Chronic liver disease
* Planned surgeries/procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Safety and Tolerability - Treatment-emergent Adverse Events | 12 weeks
  Summary of treatment emergent adverse events coded using MedDRA

SECONDARY OUTCOMES:
Evaluation of Pharmacokinetics - PK | 12 weeks
  Peak plasma concentration of SGM-1019 as measured by Cmax
Evaluation of Pharmacodynamics - Labs | 12 weeks
  Evaluation of liver functions labs of ALT, AST, ALP, and bilirubin.
Evaluation of Phamacodynamics - MRI | 12 weeks
  Evaluation of MRI parameters for assessment of liver fat, fibroinflammation, and stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W McClure, M.D., Study Director — Second Genome
Locations (10):
- United States (10):
  - Second Genome Clinical Site 405, Chandler, Arizona
  - Second Genome Clinical Site 406, Tucson, Arizona
  - Second Genome Clinical Site 403, Panorama City, California
  - Second Genome Clinical Site 409, Lakewood Rch, Florida
  - Second Genome Clinical Site 410, Flowood, Mississippi
  - Second Genome Clinical Site 404, Kansas City, Missouri
  - Second Genome Clinical Site 408, Fayetteville, North Carolina
  - Second Genome Clinical Site 407, Clarksville, Tennessee
  - Second Genome Clinical Site 402, Austin, Texas
  - Second Genome Clinical Site 401, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No